CLINICAL TRIAL: NCT03400657
Title: A Prospective, Multicenter, Prospective, Non-intervention, Controlled Trial of MDT to Evaluate the Survival Benefit of Patients With Advanced Gastric / Colorectal Cancer in Realistic Medical Practice
Brief Title: MDT to Evaluate the Survival Benefit of Patients With Advanced Gastric / Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Head of department of Gastroentestinal oncology, Peking University
Other Study IDs: CSMDT-01
Record Dates: First submitted 2018-01-02; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Multi-disciplinary Treatment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- fully implemented to the MDT decision: group of patients fully implemented to the MDT decision
  Interventions: Procedure: Multi-disciplinary Treatment
- not completly implemented to the MDT-decision: group of patients not completly implemented to the MDT decision
  Interventions: Procedure: Multi-disciplinary Treatment
- not implemented to the MDT decision: group of patients not implemented to the MDT decision
  Interventions: Procedure: Multi-disciplinary Treatment

INTERVENTIONS:
Procedure: Multi-disciplinary Treatment — due to suggestion of Multi-disciplinary Treatment ,the patients would be suggested to chemotherapy or surgery.

SUMMARY:
This is a prospective, multicenter, non-interventional, controlled clinical study. Evaluate MDT performance and benefit analysis in patients with advanced gastric or colorectal cancer after MDT discussion under real medical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological diagnosis of recurrent / metastatic gastric or colorectal cancer.
2. Participate in formal MDT discussions at the Research Center.
3. MDT decision-making at least two subjects involved in treatment.
4. Patient informed consent and signed written consent.

Exclusion Criteria:

1. Early or locally advanced gastric cancer or colorectal cancer.
2. Accept informal MDT discussions.
3. MDT decisions recommend only a single subject for treatment of patients.
4. MDT decisions recommend only palliative patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: recurrent / metastatic gastric or colorectal cancer
Sampling Method: Probability Sample
Enrollment: 484 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
overall survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

SECONDARY OUTCOMES:
Differences in overall survival after performing MDT at center | 1 years
  Differences in overall survival after performing MDT at center

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No